CLINICAL TRIAL: NCT05502536
Title: Effects of Individualized Fairytales on Preschool Children With Attention Deficit Hyperactivity Disorder With Developmental Delay
Brief Title: Effects of Fairytales on Preschool Children With Attention Deficit Hyperactivity Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022SKHADR033
Record Dates: First submitted 2022-08-14; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Developmental Delay; Preschool Children; Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Learning Disabilities; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants and outcome assessor will be blinded to the groups' allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): traditional rehabilitation programs with additional individualized fairytales class
  Interventions: Other: Traditional rehabilitation programs with Individualized fairytales class
- Control group (No Intervention): traditional rehabilitation programs without additional individualized fairytales class

INTERVENTIONS:
Other: Traditional rehabilitation programs with Individualized fairytales class — In addition to traditional rehabilitation programs, 30 minutes per week for 12 sessions of individualized fairytales classes by a child and educational teacher for three months, to preschool children with Attention Deficit Hyperactivity Disorder and developmental delays in regular traditional rehabilitation programs
  Arms: Intervention group

SUMMARY:
Under traditional rehabilitation programs, investigate the additional effects of individualized fairytales on preschool children with Attention Deficit Hyperactivity Disorder with developmental delays.

DETAILED DESCRIPTION:
Thirty preschool children with Attention Deficit Hyperactivity Disorder and developmental delays will be enrolled in regular traditional rehabilitation programs.

They will be randomized to the intervention group and control group. The participants in the intervention group will receive an additional 30 minutes per week for 12 sessions of individualized fairytales classes by a child and educational teacher for three months. The participants of both groups will continue to receive the traditional rehabilitation programs.

Therapeutic effects, including attention, cognitive function, vocabulary function, physical functional performance, and quality of life at baseline, will be evaluated after 12 weeks of treatment and three months after the treatment.

The evaluator will be blinded to the group's allocation during the whole course of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* preschool children with a diagnosis of Attention Deficit Hyperactivity Disorder and developmental delay, under regular traditional rehabilitation programs, intelligence quotient 70 or greater

Exclusion Criteria:

* age less than 3 or greater than 6 of children diagnosed with Attention Deficit Hyperactivity Disorder and developmental delay, under regular traditional rehabilitation programs, intelligence quotient below 70

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-08-20 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
changes of hyperactivity | score change from baseline to 12 weeks of treatment, and 12 weeks after treatment
  score assessed by Swanson, Nolan and Pelham questionnaire, higher score indicating greater hyperactivity
changes of attention | score change from baseline to 12 weeks of treatment, and 12 weeks after treatment
  score change by Conners Kiddie Continuous Performance Test, greater score indicating lower attention span

SECONDARY OUTCOMES:
change of vocabulary | score change from baseline to 12 weeks of treatment, and 12 weeks after treatment
  score change by Receptive and Expressive Vocabulary Test, higher score indicating greater performance
change of sensory integration | score change from baseline to 12 weeks of treatment, and 12 weeks after treatment
  score change by Sensory Profile, 0-100, higher score indicating better sensory profile
change of intelligence | score change from baseline to 12 weeks of treatment, and 12 weeks after treatment
  score change by Wechsler Intelligence Scale for Children, the average score is 100, with a higher score indicating higher intelligence and a lower score indicating a lower level of intelligence
change of physical functional performance | score change from baseline to 12 weeks of treatment, and 12 weeks after treatment
  score assessed by Pediatric Outcome Data Collection Instrument, 0-100, a higher score indicating greater performance
change of quality of life | score change from baseline to 12 weeks of treatment, and 12 weeks after treatment
  score assessed by the Pediatric Quality of Life Inventory, 0-100, a higher score indicating a greater quality of life
change of family impact | score change from baseline to 12 weeks of treatment, and 12 weeks after treatment
  score assessed by Child Health Questionnaire, parent form 28, 0-100, a higher score indicating better performance
change of walking time | score change from baseline to 12 weeks of treatment, and 12 weeks after treatment
  walking time
change of stairs climbing time | score change from baseline to 12 weeks of treatment, and 12 weeks after treatment
  climbing time
change of balance | score change from baseline to 12 weeks of treatment, and 12 weeks after treatment
  one leg standing time
change of physical function | score change from baseline to 12 weeks of treatment, and 12 weeks after treatment
  5 times sit to stand up

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Lan Hsieh, MD, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No